CLINICAL TRIAL: NCT04100772
Title: A Randomized,Blind, Positive-controlled Phase I Clinical Trial to Preliminary Evaluate the Safety and Immunogencity of 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT） in Healthy People Aged 6 Weeks and Above
Brief Title: Phase I Clinical Trial of a Candidate PCV13 in Healthy People Aged 6 Weeks and Above
Acronym: PICTPCV13i
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CS-CTP-PCV
Record Dates: First submitted 2019-09-18; First posted 2019-09-24 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Pneumococcal Infections; Streptococcal Infections; Bacterial Infections
Keywords: PCV13; 13 valent Pneumococcal conjugate vaccine; Pneumococcal Infections; Safety; Immunogenicity
MeSH Terms: conditions — Pneumococcal Infections; Streptococcal Infections; Bacterial Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- vaccine 1A (Experimental): Subjects received one dose of PCV13i at 18 to 49 years old
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT）
- vaccine 2A (Experimental): Subjects received one dose of PCV13i at 50 years old and above
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT）
- vaccine 3A (Experimental): Subjects received one dose of PCV13i at 6 to 17 years old
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT）
- vaccine 4A (Experimental): Subjects received one dose of PCV13i at 2 to 5 years old
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT）
- vaccine 5A (Experimental): Subjects received two doses of PCV13i at 7 months to 2 years old
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT）
- vaccine 6A (Experimental): Subjects received three doses of PCV13i at 3,4,5 months of age
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT）
- vaccine 7A (Experimental): Subjects received three doses of PCV13i at 2,4,6 months of age
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT）
- vaccine 7B (Active Comparator): Subjects received three doses of PCV13 at 2,4,6 months of age
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine

INTERVENTIONS:
Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT） — 0.5mL,Intramuscular other name:PCV13i
  Arms: vaccine 1A; vaccine 2A; vaccine 3A; vaccine 4A; vaccine 5A; vaccine 6A; vaccine 7A
Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine — 0.5mL,Intramuscular other name:Prevnar
  Arms: vaccine 7B

SUMMARY:
Streptococcus pneumoniae is a major cause of morbidity and mortality in children worldwide, resulting in up to 1 million pediatric deaths every year.Since the licensure of PCV7 and PCV13,the reported overall decline in invasive pneumococcal disease in hospitalized children younger than 5 years several years is approximately 60% in Western countries.This is a single center,blind, randomized, positive-controlled clinical trial.The purpose of this study is to preliminary evaluate the safety of PCV13i vaccine in subjects at age of 7 months and above,and to investigate the safety and immunogenicity of PCV13i vaccine at age of 2 and 3 months,compared to PCV13.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects of 2 months (minimum 6 weeks), 3 months , 7 months and above;
* Willing to provide proof of identity;
* Without vaccination history of pneumococcal vaccine;
* None-pregnancy or do not plan to pregnancy recently;;
* Volunteers of 18 years old and above who have the ability to understand clinical studie progress and sign informed consent;
* Volunteers of 8-17 years old and their guardians who willing sign informed consent;
* Able to understand and sign the informed consent by their guardians or trustees for the volunteers of 8 years old and below;
* Able and willing comply with the requirements of the protocol ;

Exclusion Criteria:

* Volunteers whose axillary body temperature was >37.0℃ before vaccination
* Volunteers who suffered from Congenital malformation or developmental disorder, genetic defect, severe malnutrition, etc;
* Volunteers who has a history of epilepsy, convulsions or psychosis;
* -Allergic person;
* Any prior administration of blood products in last 3 month;
* Any prior administration of other research medicines in last 1 month;
* Plans to participate in or is participating in any other drug clinical study;
* Any prior administration of attenuated live vaccine in last 14 days;
* Any prior administration of subunit or inactivated vaccines in last 7 days;
* Had fever before vaccination, Volunteers with temperature >37.0°C on axillary setting;
* According to the investigator's judgement, the subjects have any other factors that make them unfit to enroll the clinical trial

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Safety items of adverse reactions | within 7 days post each vaccination
  Occurrence of adverse reactions of each subject(Arm 1A-7B)
Safety items of SAE | within 6 months post last vaccination
  Occurrence of SAE of each subject(Arm 1A-7B)
Safety items of Hematological examination | day 4 post vaccination
  Occurrence of abnormal changes of Hematological examination in subjects of 2 years old and above(Arm 1A-4A)
Safety items of Urine test | day 4 post vaccination
  Occurrence of abnormal changes of Urine test in subjects of 2 years old and above(Arm 1A-4A)
Safety items of Blood chemistry test | day 4 post vaccination
  Occurrence of abnormal changes of Blood chemistry test in subjects of 2 years old and above(Arm 1A-4A)
Safety items of pressure value | day 4 post vaccination
  Occurrence of abnormal changes of pressure valus in subjects of 18 years old and above(Arm 1A-2A)
Safety items of heart rate | day 4 post vaccination
  Occurrence of abnormal changes of heart rate in subjects of 18 years old and above(Arm 1A-2A)
Safety items of adverse reactions | within 30 days post each vaccination
  Occurrence of adverse reactions of each subject(Arm 1A-7B)

SECONDARY OUTCOMES:
immunogencity items of seropositivity rates by ELISA | day 30 post last vaccination
  Serotype-specific seropositivity rates of Immunoglobulin G concentrations above 0.35ug/ml in subjects aged 2 and 3 months post last vaccination(Arm 6A-7B)
immunogencity items of GMC by ELISA | day 30 post last vaccination
  Serotype specific IgG GMC of each the pneumococcal serotypes in subjects aged 2 and 3 months post last vaccination(Arm 6A-7B)
immunogencity items of GMI by ELISA | day 30 post last vaccination
  Serotype-specific GMI value pneumococcfor each of the pneunococcal serotypes in subjects aged 2 and 3 months post last vaccination(Arm 6A-7B)
immunogencity items of GMT | day 30 post last vaccination
  Serological response in terms of GMT for each of the pneumococcal serotypes tested by OPA in subjects aged 2 months post last vaccination(7A、7B)

CONTACTS AND LOCATIONS:
Overall Officials: Xia Shengli, Principal Investigator — Henan Province Center for Disease Control and Prevention
Locations (1):
- Neihuang Center for Disease Control and Prevention, Anyang, Henan, China

IPD SHARING:
Plan to Share IPD: No
In order to maintain the rights of the subject, do not open the IPD